CLINICAL TRIAL: NCT03667950
Title: Vascular Border Zone Definition Using Intraoperative Hyperspectral Imaging for Resections and Reconstructions in Diseases of the Esophagus, Stomach, Pancreas, Small Intestine, Large Intestine and Rectum to Optimize Anastomotic Healing
Brief Title: Intraoperative Hyperspectral Imaging in Gastrointestinal Anastomoses
Acronym: HSIGI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Dr. Boris Jansen-Winkeln, Dr., University of Leipzig
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HSIGI
Record Dates: First submitted 2018-08-30; First posted 2018-09-12 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Surgical Anastomosis
Keywords: anastomotic perfusion, tissue oxygen saturation
MeSH Terms: interventions — Hyperspectral Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hyperspectral imaging (Experimental): diagnostic hyperspectral Imaging of the gastrointestinal anastomosis and calculating the anastomotic Perfusion measures
  Interventions: Procedure: Hyperspectral Imaging

INTERVENTIONS:
Procedure: Hyperspectral Imaging — Photos were taken with the hyperspectral camera of the gastrointestinal anastomosis.

SUMMARY:
In this study, gastrointestinal anastomoses are examined with a hyperspectral camera.

DETAILED DESCRIPTION:
The anastomoses were examined under standardized conditions directly after creation. The measurements were performed like described before, using the TIVITA Tissue system (Diaspective Vision GmbH, Am Salzhaff, Germany). This HSI-camera provides hyperspectral images with a high spectral resolution (5 nm) in the visible and near infrared range (500-1000 nm). The distance between camera and object was 30 cm for all measurements. The Number of Effective Pixels at this distance is 640 × 480 (x-, y-axis. The resulting field of view (FOV) has the dimensions 6.4 × 4.8 cm2 and a spatial resolution of 0.1 mm/pixel. The FOV is illuminated by 8 halogen spots (20 W each). The ceiling lights and other light sources were switched off, to avoid artifacts during the measurement (approximately 10 seconds). A RGB image and 4 false color images that represent physiologic parameters are intraoperatively provided by an analysis software. This work is focused on tissue oxygenation (StO2), which represents the relative blood oxygenation in the microcirculation of superficial tissue layers (approximately 1 mm) and the near-infrared (NIR) Perfusion Index, representing tissue layers in 4-6 mm penetration depth.

ELIGIBILITY:
Inclusion Criteria:

* all gastrointestinal anastomoses

Exclusion Criteria:

* inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Anastomotic Perfusion: (Oxygenation (StO2) | direct during the Operation (ca. 15-20 Minutes)
  Oxygenation (StO2) in %: Relative O2 saturation of the blood immicrocircular system in superficial tissue layers (penetration depth: approx. 1 mm)
Anastomotic Perfusion: Tissue-Hemoglobin index | direct during the Operation (ca. 15-20 Minutes)
  Tissue Hemoglobin index in %: Existing hemoglobin distribution in the microcircular system of the tissue area under consideration (index value)
Anastomotic Perfusion: Near Infrared Perfusion Index | direct during the Operation (ca. 15-20 Minutes)
  Near Infrared Perfusion Index in %: Relative O2 saturation of the blood immicrocircular system in deeper tissue layers (penetration depth: 4-6mm; index value)
Anastomotic Perfusion: Tissue-Water-Index | direct during the Operation (ca. 15-20 Minutes)
  Tissue-Water-Index in %: Existing water distribution in the tissue area under consideration (index value)

CONTACTS AND LOCATIONS:
Overall Officials: Boris Jansen-Winkeln, Dr., Principal Investigator — University of Leipzig
Locations (1):
- Universitätsklinikum Leipzig - AöR, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No
no sharing

REFERENCES:
- [Background] Jansen-Winkeln B, Maktabi M, Takoh JP, Rabe SM, Barberio M, Kohler H, Neumuth T, Melzer A, Chalopin C, Gockel I. [Hyperspectral imaging of gastrointestinal anastomoses]. Chirurg. 2018 Sep;89(9):717-725. doi: 10.1007/s00104-018-0633-2. German. PMID 29637244